CLINICAL TRIAL: NCT04608955
Title: A Multi-center, Randomized, Positive-controlled Phase 2 Clinical Trial to Evaluate the Early Bactericidal Activity, Safety and Tolerability of WX-081 in Participants With Drug-naive&Susceptible or Drug-Resistant Pulmonary Tuberculosis
Brief Title: Evaluation of Early Bactericidal Activity and Safety in Pulmonary Tuberculosis With WX-081
Acronym: WX-081
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiatan Pharmatech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JYB0201
Record Dates: First submitted 2020-10-10; First posted 2020-10-30 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Tuberculosis
Keywords: Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — sudapyridine; bedaquiline

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Arm A: WX-081 (Experimental): Participants with newly-treated drug sensitivity tuberculosis receive WX-081 150mg orally once daily for 2 weeks.
  Interventions: Drug: WX-081
- Arm B: WX-081 (Experimental): Participants with newly-treated drug sensitivity tuberculosis receive WX-081 300mg orally once daily for 2 weeks.
  Interventions: Drug: WX-081
- Arm C: WX-081 (Experimental): Participants with newly-treated drug sensitivity tuberculosis receive WX-081 450mg orally once daily for 2 weeks.
  Interventions: Drug: WX-081
- Arm D: Standard treatment (Active Comparator): Participants with newly-treated drug sensitivity tuberculosis receive standard treatment for two weeks.
  Interventions: Drug: Standard treatment
- Arm E: WX-081+MBT (Experimental): Participants with drug-resistant tuberculosis receive WX-081 400mg orally once daily for 2 weeks, and then MBT+ WX-081 150mg orally once daily for 6 weeks.
  Interventions: Drug: WX-081; Drug: Multi-drug background treatment (MBT)
- Arm F: Bedaquiline+MBT (Active Comparator): Participants with drug-resistant tuberculosis receive Bedaquiline 400mg orally once daily for 2 weeks, and then MBT+ Bedaquiline 200mg orally 3 times per week for 6 weeks.
  Interventions: Drug: Bedaquiline; Drug: Multi-drug background treatment (MBT)

INTERVENTIONS:
Drug: WX-081 — WX-081 is not licensed yet. WX-081 will be used in arms A, B, C, WX-081+MBT.
  Arms: Arm A: WX-081; Arm B: WX-081; Arm C: WX-081; Arm E: WX-081+MBT
Drug: Bedaquiline — This licensed drug will be used in arm F as positive comparator.
  Arms: Arm F: Bedaquiline+MBT
Drug: Standard treatment — Standard treatment will be used in arm D as positive comparator, according to the recommendations of WHO guidelines for diagnosis and treatment of tuberculosis.
  Arms: Arm D: Standard treatment
Drug: Multi-drug background treatment (MBT) — MBT will be used in arm E, F as background treatment. The drugs used in MBT are all licensed drugs, and the treatment complies with the recommendations of WHO guidelines for diagnosis and treatment of tuberculosis.
  Arms: Arm E: WX-081+MBT; Arm F: Bedaquiline+MBT

SUMMARY:
This is a multi-center, randomized, parallel, open-label, positive-controlled Phase 2 clinical trial, which aims to evaluate the early bactericidal activity, safety and tolerability of WX-081 in patients with drug-naive&susceptible and drug-resistant tuberculosis. Also the efficacy of WX-081 will be explored in participants with drug-resistant tuberculosis.

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, randomized, parallel, open-label, positive-controlled clinical trial. The objective of this trial is to evaluate the early bactericidal activity, safety and tolerability of WX-081 patients with drug-naive&susceptible and drug-resistant tuberculosis. and the efficacy in participants with drug-resistant tuberculosis.

This trial will be divided into core research stage (stage 1) and extended research stage (stage 2). During stage 1, a panel of 59 participants with drug-naive&susceptible tuberculosis will be randomized to receive either WX-081(including 3 groups:150mg qd, 300mg qd, 450mg qd. n=12 per group) or standard treatment (n=8) for 2 weeks, and then followed by a follow-up period of 2 weeks. A panel of 40 participants with drug-resistant tuberculosis will be randomized to receive either WX-081 (400mg qd, n=20) or bedaquiline (400mg qd, n=20) for 2 weeks. During stage 2, the 40 participants with drug-resistant tuberculosis will receive WX-081(150mg qd) + MBT treatment (ie. multi-drug background treatment) and bedaquiline (200mg tiw) +MBT treatment for 6 weeks respectively, and then followed by a follow-up period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged between 18 and 65 years.
2. Body weight between 40 and 90 kg.
3. Newly-treated drug sensitivity tuberculosis: clinically diagnosed as pulmonary tuberculosis, without treatment, sputum smear-positive for acid-fast bacilli (AFB at least 1+), and no resistant to rifampicin or isoniazid in the drug sensitivity test.
4. Drug-resistant tuberculosis: re-treatment pulmonary tuberculosis patients, diagnosed as rifampicin resistance (RR-TB) or isoniazid and rifampicin resistance (MDR-TB) by molecular biology methods, and sputum smear-positive for acid-fast bacilli. Patients must be willing to discontinue all TB drugs to allow 7 days washout.
5. Patients must consent to HIV-testing, or provide HIV-negative report within 6 months.
6. Women are not breastfeeding or pregnant, and agree to practice effective contraception throughout the trial.
7. Provide voluntary and written informed consent prior to all trial-related procedures, agree to comply with the requirements and restrictions listed in the informed consent form and agreement.

Exclusion Criteria:

1. Patients with HIV infection.
2. Patients with miliary tuberculosis or extrapulmonary tuberculosis judged by the investigator.
3. Patients with certain QT/QTc interval characteristics as described in the protocol.
4. the patients have a history of, or current evidence of clinically relevant unstable or severe cardiovascular, kidney, liver, blood, tumor, endocrine and metabolic, mental or rheumatic diseases, or any other condition that will not be suitable to participate in this study, according to the judgement of the investigator.
5. Patients who have participated in other clinical studies within 8 weeks prior to trial start.
6. Patients having a known or suspected hypersensitivity or serious adverse reaction to drugs used in this trial.
7. Women who are pregnant, breastfeeding, or planning to become pregnant.
8. Current or past history of alcohol and/or drug use that, in the investigator's opinion, would compromise the participant's safety or compliance to the study protocol procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Time to positive (TTP) | Day 0-14.
  TTP is measured as time to sputum culture positivity in Liquid Culture Media.
Early bactericidal activity (EBA) of WX-081 | Day 0-14.
  EBA is measured as the mean rate of colony forming unit (log10CFU) of mycobacterium tuberculosis per ml sputum on solid medium in different time periods.

SECONDARY OUTCOMES:
change of electrocardiogram QT interval | Measured through 8 Weeks.
  QT interval is calculated as QTcF in milliseconds (ms)
The percentage of participants with sputum culture-negative conversion. | Measured through 8 Weeks.
  Percentage of participants with an occurrence of sputum culture-negative through 8 weeks.
Rate of change of colony forming units (CFU) | Measured through 8 Weeks.
  Rate of change of colony forming units (CFU) of mycobacterium tuberculosis on sputum culture through 8 weeks.
The percentage of participants with sputum smear-negative conversion. | Measured through 8 Weeks.
  Percentage of participants with an occurrence of sputum smear-negative through 8 weeks.
heart rate | Measured through 8 Weeks.
  heart rate in times per minute.
blood pressure | Measured through 8 Weeks.
  blood pressure in mmHg
Maximum plasma concentration (Cmax) | At day1 and 14.
  Blood samples will be taken at different time points before and after administration on Day1 and Day14 of treatment.
Time to reach maximum plasma concentration (Tmax) | At day1 and 14.
  Blood samples will be taken at different time points before and after administration on Day1 and Day14 of treatment.
Area under the plasma concentration versus time curve (AUC(0-t)) | At day1 and 14.
  Blood samples will be taken at different time points before and after administration on Day1 and Day14 of treatment.
Terminal plasma half-life (t1/2) | At day1 and 14.
  Blood samples will be taken at different time points before and after administration on Day1 and Day14 of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Song AiYun, MD, Study Chair — Shang hai Jiatan Pharma
Locations (1):
- Beijing Chest Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang Z, Luo W, Xu D, Guo F, Yang M, Zhu Y, Shen L, Chen S, Tang D, Li L, Li Y, Wang B, Franzblau SG, Ding CZ. Discovery and preclinical profile of sudapyridine (WX-081), a novel anti-tuberculosis agent. Bioorg Med Chem Lett. 2022 Sep 1;71:128824. doi: 10.1016/j.bmcl.2022.128824. Epub 2022 May 27. PMID 35636648